CLINICAL TRIAL: NCT03153891
Title: Virtual Nature: Benefits for Older Adults Who Experience Chronic Pain?
Brief Title: Nature as a Buffer Among People With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1703006971
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Chronic Pain
Keywords: environment; nature
MeSH Terms: conditions — Chronic Pain | interventions — Built Environment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Natural Environment (Experimental): Participants experience a virtual reality natural environment intervention (using VR goggles with Smartphone) for 10 minutes on two occasions, 1 week apart.
  Interventions: Other: Natural Environment
- Built Environment (Experimental): Participants experience a virtual reality built environment intervention (using VR goggles with Smartphone) for 10 minutes on two occasions, 1 week apart.
  Interventions: Other: Built Environment
- Control (No Intervention): Participants do not experience a VR intervention. Instead they visit with research assistants for 10 minutes on two occasions, 1 week apart.

INTERVENTIONS:
Other: Natural Environment — the natural environment will be delivered via Samsung VR gear goggles with Samsung smartphone.
  Other Names: VR nature
  Arms: Natural Environment
Other: Built Environment — the built environment will be delivered via Samsung VR gear goggles with Samsung smartphone.
  Other Names: VR built environment
  Arms: Built Environment

SUMMARY:
This randomized controlled trial examines the effect of nature exposure on pain intensity levels among older adults who experience chronic pain. Investigators examine the effects of nature on: the experience of chronic pain, on pain catastrophizing, and on attention restoration.

DETAILED DESCRIPTION:
Nature has been used to reduce pain in the context of acute pain (e.g., during painful medical procedures) but nature has not been examined as an intervention strategy to address chronic pain. Second, the mechanism though which nature might reduce the experience of pain is not well understood. Participants are cognitively intact individuals aged 60-90 who experience chronic pain and who rate their health as fair, good or excellent. Participants are randomly assigned to one of three conditions: virtual reality (VR) nature; VR built environment; or control. Researchers examine effects of VR nature exposure on the experience of chronic pain, pain catastrophizing, and on attention restoration as well as the relations among these variables.

ELIGIBILITY:
Inclusion Criteria:

* rate health as "fair" "good" or "excellent"
* experience chronic pain
* cognitively intact
* do not use wheelchair

Exclusion Criteria:

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Experience of chronic pain | up to 3 weeks; from date of randomization until 2nd data collection date
  rating of pain intensity, on scale of 1-10

SECONDARY OUTCOMES:
Pain catastrophizing | up to 3 weeks; from date of randomization until 2nd data collection date
  rate 13 items on 5-point scale (0-4) (Sullivan, et al., 2001)
cognitive functioning | up to 3 weeks; from date of randomization until 2nd data collection date
  attention restoration - digit span forward & backwards; Attention Network Test

CONTACTS AND LOCATIONS:
Overall Officials: Nancy M Wells, PhD, Principal Investigator — Design + Environmental Analysis, Cornell University
Locations (1):
- Cornell University, Ithaca, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to share individual participant data with other researchers.